CLINICAL TRIAL: NCT01228799
Title: Longterm Comparison Between Trabeculectomy and Canaloplasty in Open-angle Glaucoma
Brief Title: Trabeculectomy Versus Canaloplasty
Acronym: TVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Eye Hospital, Würzburg (Other)
Responsible Party: University Eye Hospital, University Hospitals Würzburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TVC-1; TVC (Other: University Eye Hospital Wurzburg)
Record Dates: First submitted 2010-10-20; First posted 2010-10-27 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2010-10

CONDITIONS: Glaucoma; Canaloplasty; Trabeculectomy
Keywords: trabeculectomy,; canaloplasty,; glaucoma surgery; non-penetrating surgery
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trabeculectomy (Active Comparator): Trabeculectomy with Mitomycin C
  Interventions: Procedure: trabeculectomy
- Canaloplasty (Active Comparator): Canaloplasty with implant of suture
  Interventions: Procedure: Canaloplasty

INTERVENTIONS:
Procedure: trabeculectomy — trabeculectomy with mitomycin C 0.2mg/ml
  Arms: Trabeculectomy
Procedure: Canaloplasty — Canaloplasty with implant of suture
  Arms: Canaloplasty

SUMMARY:
Study aims for comparison of trabeculectomy and canaloplasty, in order to find out if one operation is superior to the other. Both procedures are performed in patients with medically uncontrolled open-angle glaucoma. Canaloplasty is a recently newly introduced procedure, which showed encouraging results without antimetabolite usage intra- and postoperatively. Purpose of the study is to compare both surgeries concerning success rate, intraocular pressure, medication and complications. So far there is no comparison of the standard procedure trabeculectomy and the new approach, canaloplasty available.

ELIGIBILITY:
Inclusion Criteria:1. diagnosed primary or secondary open-angle glaucoma 2. IOP > 16 mmHg (<60 days prior surgery) 3. IOP > 21 mmHg 4. no prior glaucoma surgery (once laser trabeculoplasty or cyclophotocoagulation) allowed

Exclusion Criteria:

1. angle closure glaucoma
2. congenital glaucoma
3. combined procedures (glaucoma and cataract)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
success rate (complete and qualified success) | 1 year
  Success is defined 1. IOP < 21 mmHg and at least 20% IOP reduction from baseline 2. IOP < 18 mmHg
success rate (complete and qualified success) | 2 years
  Success is defined 1. IOP < 21 mmHg and at least 20% IOP reduction from baseline 2. IOP < 18 mmHg

SECONDARY OUTCOMES:
IOP, medication, complications | 1 year
  intraocular pressure reduction, medication postoperatively, complications intra- and postoperatively
IOP, medication, complications | 2 years
  intraocular pressure reduction, medication postoperatively, complications intra- and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klink, MD, Principal Investigator — University Eye Hospital, Würzburg
Locations (1):
- University Eye Hospital, Würzburg, Bavaria, Germany